CLINICAL TRIAL: NCT01747915
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP, MULTI-CENTER TRIAL OF PREGABALIN AS ADJUNCTIVE THERAPY IN PEDIATRIC AND ADULT SUBJECTS WITH PRIMARY GENERALIZED TONIC-CLONIC SEIZURES - PROTOCOL A0081105
Brief Title: A Safety, Efficacy and Tolerability Trial of Pregabalin as Add-On Treatment in Pediatric and Adult Subjects With Primary Generalized Tonic-Clonic (i.e., Grand Mal) Seizures.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081105; 2010-023263-18 (EudraCT Number)
Record Dates: First submitted 2012-11-27; First posted 2012-12-12 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2019-08

CONDITIONS: Generalized Tonic Clonic Seizures
Keywords: Primary Generalized Tonic Clonic Seizures; Epilepsy; Safety; Efficacy; Tolerability; Pregabalin; Lyrica; Adjunctive treatment; Placebo Controlled; Blinded
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study Drug Level 1 (Experimental)
  Interventions: Drug: Pregabalin Dose Level 1
- Study Drug Level 2 (Experimental)
  Interventions: Drug: Pregabalin Dose Level 2
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin Dose Level 1 — Pregabalin, either liquid or capsule, dosed twice daily, escalated up to a maximum of 300 mg/day beginning at Randomization to Taper Phase, then tapered down to a maximum dose of 150 mg/day during 1 week Taper Phase to End of Study/Early Termination.
  Other Names: Lyrica Dose Level 1
  Arms: Study Drug Level 1
Drug: Pregabalin Dose Level 2 — Pregabalin, either liquid or capsule, dosed twice daily, escalated up to a maximum of 600 mg/day beginning at Randomization to Taper Phase, then tapered down to a maximum of 150 mg/day during 1 week Taper Phase to End of Study/Early Termination.
  Other Names: Lyrica Dose Level 2
  Arms: Study Drug Level 2
Drug: Placebo — Placebo, either liquid or capsule, dosed twice daily beginning at Randomization to End of Study/Early Termination.
  Arms: Placebo

SUMMARY:
The study is designed to evaluate the safety, tolerability and efficacy of two doses of pregabalin as add-on treatment in pediatric and adult subjects with Primary Generalized Tonic-Clonic (PGTC) seizures as compared to placebo. It is hypothesized that both doses of pregabalin will demonstrated superior efficacy when compared to placebo by reducing PGTC seizure frequency and that pregabalin will be safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Seizures classified as Primary Generalized Tonic Clonic Seizures
* Must have at least 1 PGTC seizure in the 8 weeks prior to screening
* Must have a minimum of 3 PGTC seizures during the 8-week baseline phase and at least 1 PGTC in each 4-week period of the baseline phase
* Currently receiving adequate and stable dosage of 1 to 3 anti-epileptic treatments (stable within 28 days of screening)
* Signed informed consent and assent if a minor
* Ability to comply with daily seizure and dosing diary requirements and all study procedures

Exclusion Criteria:

* A current diagnosis of febrile seizures, or seizures related to an ongoing acute medical illness
* Focal seizures (simple partial, complex partial, or partial becoming secondarily generalized)
* Status Epilepticus within 1 year prior to screening
* Lennox-Gastaut syndrome, infantile spasms, Benign Epilepsy with Centrotemporal Spikes (BECTS) and Dravet syndrome
* Seizures related to drugs, alcohol, or acute medical illness
* Any change in anti-epileptic treatment regimen (type of medication or dose; VNS alteration) within 28 days of the screening visit or during the baseline phase
* Progressive or potentially progressive structural CNS lesion or a progressive encephalopathy.
* Progressive inborn errors of metabolism.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2013-04-03 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (124):
- United States (12):
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - Pediatric Epilepsy Center of Central Florida, Orlando, Florida
  - Pediatric Neurology, PA, Orlando, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Chinmay K. Patel, D.O., Hoffman Estates, Illinois
  - St. Alexius Medical Center, Hoffman Estates, Illinois
  - Ohio Clinical Research Partners, LLC, Canton, Ohio
  - Road Runner Research, Ltd, San Antonio, Texas
  - Scott & White Memorial Hospital and Clinic, Temple, Texas
  - Rainier Clinical Research Center, Inc., Renton, Washington
- Austria (2):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - AKH Linz, Linz
- UZ Vitebsk Regional Childrens Clinical Centre, Vitebsk, Belarus
- Bosnia and Herzegovina (4):
  - University Clinical Center Sarajevo, Sarajevo, Canton Sarajevo
  - University Clinical Center Tuzla, Tuzla, Canton Tuzla
  - University Clinical Hospital Mostar, Mostar, Herzegovinaneretva Canton
  - Public Health Institution Hospital Dr Mladen Stojanovic, Prijedor, Republika Srpska
- Bulgaria (8):
  - Multiprofile Hospital for Active Treatment Puls AD, Blagoevgrad
  - DCC Sv. Pantaleimon OOD, Pleven
  - Military Medical Academy - Multiprofile Hospital for Active Treatment, Pleven
  - MHAT Central Onco Hospital OOD, Plovdiv
  - Medical Center Teodora, Rousse
  - MHATNP Sveti Naum EAD, Sofia
  - UMHAT Aleksandrovska, Sofia
  - DCC Sveta Anna - Sofia, Sofia
- China (3):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shanghai Huashan Hospital, Neurology Department, Shanghai, Shanghai Municipality
- University Hospital Center Split, Clinic for Neurology, Split, Croatia
- Denmark (2):
  - Aarhus University Hospital, Aarhus C
  - Odense University Hospital, Odense C
- France (3):
  - CHU d'Amiens - Picardie, Amiens
  - CHRU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU d'Amiens Hopital Pontchaillou, Rennes
- Greece (4):
  - Eginition Hospital, Athens
  - Athens Medical Center, Athens
  - General Children's Hospital Penteli, Athens
  - University General Hospital of Thessaloniki "AHEPA", Thessaloniki
- Hungary (3):
  - Semmelweis Egyetem, I. Sz. Gyermekgyogyaszati Klinika, Budapest
  - Csongrad Megyei Egeszsegugyi Ellato Kozpont Hodmezovasarhely-Mako, Hódmezővásárhely
  - Pest Megyei Flór Ferenc Kórhaz, Kistarcsa
- India (7):
  - St. John's Medical College Hospital, Bangalore, Karnataka
  - Mangala Hospital & Mangala Kidney Foundation, Mangalore, Karnataka
  - P D Hinduja National Hospital and Medical Research Centre, Mumbai, Maharashtra
  - Getwell Hospital and Research Institute, Nagpur, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - KEM Hospital Research Centre, Pune, Maharashtra
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
- Lebanon (2):
  - Saint George Hospital - University Medical Center, Beirut
  - Ain Wazein Medical Village, El Chouf
- Hospital Raja Permaisuri Bainun, Ipoh, Perak, Malaysia
- Pzu Neuron, Bijelo Polje, Montenegro
- Philippines (7):
  - Cebu Doctors' University Hospital, Cebu City, CEBU
  - Perpetual Succour Hospital, Cebu City, CEBU
  - Cebu Doctors' University Hospital, Rm Ph 7, Cebu City
  - Manila Doctors Hospital, Manila
  - Metropolitan Medical Center, Manila
  - University of Santo Tomas Hospital, Manila
  - St. Luke's Medical Center Cathedral Heights Building, Quezon City
- Poland (9):
  - COPERNICUS Podmiot Leczniczy Spzoo, Gdansk
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Katowice
  - NZOZ Novo Med, Katowice
  - Neuro-Care Gabriela Klodowska, Katowice
  - NZOZ "HIPOKRATES II" Sp. z o.o., Krakow
  - Instytut Medycyny Wsi im. Witolda Chodzki w Lublinie, Lublin
  - Solumed Centrum Medyczne, Poznan
  - NZOZ IGNIS dr n. med. Alicja Lobinska, Świdnik
  - Lecznica Medyczna ''Zycie", Warsaw
- Romania (6):
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed, Brasov
  - CMI Neurologie, Neurofiziologie (EEG, EMG, PEC) Roceanu Adina Maria, Bucharest
  - Sapiens Medical Center, Bucharest
  - Spitalul Clinic de Urgenta "Prof. Dr. Nicolae Oblu", Iași
  - Spitalul Clinic de Urgente pentru Copii "Sf. Maria", Iași
  - Spitalul de Psihiatrie "Dr. Gh. Preda", Sibiu
- Russia (18):
  - SPHI Leningrad Regional Psychoneurological Dispensary, Pgt. Roshchino, Leningradskaya Oblast'
  - Nizhmedklinika, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Perm State Medical University n. a. acad. E.A. Vagner, Perm, Permskiy KRAY
  - State Budgetary Healthcare Institution of Stavropol region, Pyatigorsk, Stavropol Kray
  - GBOU VPO "Kazan State Medical University" of Roszdrav, Kazan', Tatarstan Republic
  - Republican clinical hospital, Kazan', Tatarstan Republic
  - TSBHI City Hospital No. 5 of Barnaul, Barnaul
  - MAHI of the Order of the Red Banner of Labor City Clinical Hospital No. 1, Chelyabinsk
  - Non-state Healthcare Institution, Moscow
  - LLC City Neurological Center "Sibneiromed", Novosibirsk
  - Perm State Medical University n. a. acad. E.A. Vagner, Perm
  - SPHI Leningrad Regional Psychoneurological Dispensary, Saint Petersburg
  - FSBI V.M. Bekhterev National Research Medical Center for, Saint Petersburg
  - SBHI of Saint Petersburg Psychoneurological Dispensary #5, Saint Petersburg
  - Regional State Budgetary Institution of Ministry of Health, Smolensk
  - RSBHI Smolensk Regional Clinical Hospital, Smolensk
  - GBOU VPO Smolensk State Medical University, Smolensk
  - SHI "Central Clinical Medical Unit, Ulyanovsk
- Serbia (4):
  - Institute for Child and Youth Healthcare of Vojvodina, Novi Sad, Vojvodina
  - Institute for Mental Health, Belgrade
  - University Children's Hospital, Belgrade
  - Clinical Center Kragujevac, Kragujevac
- Slovakia (2):
  - Nemocnica s poliklinikou Hlohovec, s.r.o., Hlohovec
  - Neurologicka ambulancia MUDr. Eva Gasparova, Hlohovec
- South Korea (4):
  - Keimyung University Dongsan Hospital, Daegu, Korea
  - Seoul National University Hospital, Seoul
  - Konkuk University medical center, Seoul
  - Samsung Medical Center, Seoul
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain
- Turkey (Türkiye) (4):
  - Marmara University Pendik Training and Research Hospital, Istanbul, UST Kaynarca/pendik
  - Eskisehir Osmangazi University Medical Faculty Department Of Neurology, Eskişehir
  - Dokuz Eylul Ün. Tip Fakültesi İç Hastalıkları, Izmir
  - Celal Bayar University School of Medicine, Neurology Department, Manisa
- Ukraine (11):
  - Komunalna ustanova "Odeska oblasna psykhiatrychna likarnia 2", S. Oleksandrivka, Komintern. R-N, Odeska OBL.
  - Komunalnyi zaklad "Dnipropetrovska dytiacha miska klinichna likarnia No. 5", Dnipro
  - Komunalnyi zaklad "Dnipropetrovska oblasna dytiacha klinichna likarnia", Dnipro
  - Ivano-Frankivska oblasna dytiacha klinichna likarnia, Ivano-Frankivsk
  - Derzhavna ustanova "Instytut nevrolohii, psykhiatrii ta narkolohii, Kharkiv
  - Komunalne nekomertsiine pidpryiemstvo Kharkivskoi oblasnoi rady "Oblasna klinichna psykhiatrychna li, Kharkiv
  - Derzhavnyi zaklad "Ukrainskyi medychnyi tsentr reabilitatsii ditei z, Kyiv
  - Komunalnyi zaklad Lvivskoi oblasnoi rady "Lvivska oblasna klinichna likarnia", Lviv
  - Komunalne nekomertsiine pidpryiemstvo "Odeskyi oblasnyi, Odesa
  - Oblasnyi klinichnyi tsentr neirokhirurhii ta nevrolohii,, Uzhhorod
  - Komunalna ustanova "Miska klinichna likarnia #2", nevrolohichne viddilennia, Zaporizhzhia
- United Kingdom (4):
  - The Barberry National Centre for Mental Health, Birmingham, WEST Midlands
  - Barts Health NHS Foundation Trust, The Royal London Hospital, London
  - Salford Royal NHS Foundation Trust, Salford
  - ABMU Local Health Board, Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Driscoll J, Almas M, Gregorian G, Kyrychenko A, Makedonska I, Liu J, Patrick J, Scavone JM, Antinew J; 1105 Study Group. Pregabalin as adjunctive therapy in adult and pediatric patients with generalized tonic-clonic seizures: A randomized, placebo-controlled trial. Epilepsia Open. 2021 Jun;6(2):381-393. doi: 10.1002/epi4.12492. Epub 2021 May 16. PMID 34033265
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081105&StudyName=A%20Safety%2C%20Efficacy%20and%20Tolerability%20Trial%20of%20Pregabalin%20as%20Add-On%20Treatment%20in%20Pediatric%20and%20Adult%20Subjects%20with%20Primary%20Generalized%20T

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted at multiple sites in 21 countries in 219 participants between 03 April 2013 and 20 February 2019.
Groups:
- Pregabalin 5 mg/kg/Day or 7 mg/kg/Day or 300 mg/Day: Participants aged less than (<) 17 years received Pregabalin, orally, twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks in following manner: 1) body weight greater than or equal to (>=)30 kg: Pregabalin 5 milligram per kilogram per day (mg/kg/day) as capsule or oral solution (using oral solution of strength 20 milligram per milliliter [mg/mL]), up to a maximum of 300 milligram per day (mg/day); 2) body weight <30 kg: pregabalin 7 mg/kg/day as oral solution (using oral solution of strength 20 mg/mL), up to a maximum of 300 mg/day. Participants aged >=17 years received Pregabalin 300 mg/day, capsule or oral solution, orally twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks.
- Pregabalin 10 mg/kg/Day or 14 mg/kg/Day or 600 mg/Day: Participants aged <17 years received Pregabalin, orally, twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks in following manner: 1) body weight >=30 kg: Pregabalin 10 mg/kg/day as capsule or oral solution (using oral solution of strength 20 mg/mL), up to a maximum of 600 mg/day; 2) body weight <30 kg: pregabalin 14 mg/kg/day as oral solution (using oral solution of strength 20 mg/mL), up to a maximum of 600 mg/day. Participants aged >=17 years received Pregabalin 600 mg/day, capsule or oral solution, orally twice daily in equally divided doses, for the double-blind treatment phase of 12 weeks.
- Placebo: Participants aged <17 years received placebo matched to Pregabalin, orally, twice daily for the double-blind treatment phase of 12 weeks (in the form of solution for <30 kg participants; in the form of capsule or liquid oral solution for >=30 kg participants). Participants aged >=17 years received placebo matched to Pregabalin, in the form of capsule or liquid oral solution, orally, twice daily for the double-blind treatment phase of 12 weeks.
Period: Overall Study
Arm/Group | Pregabalin 5 mg/kg/Day or 7 mg/kg/Day or 300 mg/Day | Pregabalin 10 mg/kg/Day or 14 mg/kg/Day or 600 mg/Day | Placebo
Started | 75 | 72 | 72
Completed | 60 | 61 | 66
Not Completed | 15 | 11 | 6
Not completed — Other | 1 | 1 | 1
Not completed — Adverse Event | 8 | 5 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized participants who took at least 1 dose of investigational product during the double-blind treatment phase, have a baseline value and at least 1 post-baseline efficacy assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin 5 mg/kg/Day or 7 mg/kg/Day or 300 mg/Day | Pregabalin 10 mg/kg/Day or 14 mg/kg/Day or 600 mg/Day | Placebo | Total
Number analyzed (Participants) | 75 | 72 | 72 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (13.3) | 25.4 (12.7) | 26.2 (13.2) | 25.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 39 | 40 | 121
  Male | 33 | 33 | 32 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 8 | 6 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 67 | 64 | 65 | 196
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Log-transformed (Log) 28-day Seizure Rate for All Primary Generalized Tonic-Clonic (PGTC) Seizures During 12-Week Double-Blind Treatment Phase
Description: All PGTC seizures experienced during treatment phase were recorded by the participants or their parents/legal guardian in a daily seizure diary. 28-day seizure rate for all PGTC seizures= ([number of seizures in the double blind treatment phase] divided by [number of days in double blind treatment phase minus {-} number of missing diary days in treatment phase])*28. For log-transformation, the quantity 1 was added to the 28-day seizure rate for all participants to account for any possible "0" seizure incidence. This resulted in final calculation as: log transformed (28-day seizure rate +1).
Time Frame: Day 1 up to Week 12
Population: ITT population included all randomized participants who took at least 1 dose of investigational product during the double-blind treatment phase, have a baseline value and at least 1 post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Seizure per 28 days
Arm/Group | Pregabalin 5 mg/kg/Day or 7 mg/kg/Day or 300 mg/Day | Pregabalin 10 mg/kg/Day or 14 mg/kg/Day or 600 mg/Day | Placebo
Number analyzed (Participants) | 75 | 72 | 72
Seizure per 28 days | 1.17 (0.097) | 1.13 (0.095) | 1.14 (0.098)
Statistical Analysis 1: Comparison: Pregabalin 5 mg/kg/Day or 7 mg/kg/Day or 300 mg/Day vs Placebo; Estimates and p-values from an ANCOVA model including fixed effects for log transformed baseline value, region, age strata, and treatment group; Test type: Superiority; p = 0.8121, ANCOVA; Least Square (LS) Mean Difference = 0.02, 95% CI 2-sided [-0.15 to 0.19], Standard Error of Mean 0.088
Statistical Analysis 2: Comparison: Pregabalin 10 mg/kg/Day or 14 mg/kg/Day or 600 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8889, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.19 to 0.16], Standard Error of Mean 0.088

2. Secondary Outcome: Percentage of Participants With at Least 50 Percent (%) or Greater Reduction From Baseline in 28-day Primary Generalized Tonic-clonic (PGTC) Seizure Rate During the 12-Week Double-blind Treatment Phase
Description: Percentage of participants with 50% or greater reduction from baseline in 28-day seizure rate during the 12 week double blind treatment phase were reported. 28-day seizure rate for all PGTC seizures= ([number of seizures in the double blind treatment phase] divided by [number of days in double blind treatment phase minus {-} number of missing diary days in treatment phase])*28.
Time Frame: Day 1 up to Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 5 mg/kg/Day or 7 mg/kg/Day or 300 mg/Day | Pregabalin 10 mg/kg/Day or 14 mg/kg/Day or 600 mg/Day | Placebo
Number analyzed (Participants) | 75 | 72 | 72
percentage of participants | 41.3 | 38.9 | 41.7
Statistical Analysis 1: Comparison: Pregabalin 5 mg/kg/Day or 7 mg/kg/Day or 300 mg/Day vs Placebo; Test type: Superiority; p = 0.7973, Regression, Logistic — P-values were from a Logistic Regression Model including fixed effects for region, age strata and treatment; Odds Ratio (OR) = 1.095, 95% CI 2-sided [0.548 to 2.186]
Statistical Analysis 2: Comparison: Pregabalin 10 mg/kg/Day or 14 mg/kg/Day or 600 mg/Day vs Placebo; Test type: Superiority; p = 0.8474, Regression, Logistic — P-values were from a Logistic Regression Model including fixed effects for region, age strata and treatment; Odds Ratio (OR) = 0.934, 95% CI 2-sided [0.465 to 1.877]

ADVERSE EVENTS:
Time Frame: Day 1 up to end of study (Week 13)
Description: Same event may appear as adverse event (AE) and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Pregabalin 5 mg/kg/Day or 7 mg/kg/Day or 300 mg/Day | Pregabalin 10 mg/kg/Day or 14 mg/kg/Day or 600 mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/72 | 1/72
Serious Adverse Events (participants affected / at risk) | 2/75 | 2/72 | 3/72
Other Adverse Events (participants affected / at risk) | 39/75 | 41/72 | 36/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 5 mg/kg/Day or 7 mg/kg/Day or 300 mg/Day (N=75) | Pregabalin 10 mg/kg/Day or 14 mg/kg/Day or 600 mg/Day (N=72) | Placebo (N=72)
Sudden unexplained death in epilepsy (General disorders) | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 2 | 0
Seizure (Nervous system disorders) | 0 | 0 | 2
Status epilepticus (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 5 mg/kg/Day or 7 mg/kg/Day or 300 mg/Day (N=75) | Pregabalin 10 mg/kg/Day or 14 mg/kg/Day or 600 mg/Day (N=72) | Placebo (N=72)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 2 | 1
Diplopia (Eye disorders) | 1 | 1 | 1
Eye disorder (Eye disorders) | 1 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 5 | 3 | 3
Influenza like illness (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2
Sluggishness (General disorders) | 1 | 0 | 0
Therapeutic response unexpected (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral rhinitis (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 3
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Platelet count increased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 7 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 13 | 12 | 5
Dysgraphia (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Head titubation (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 7 | 11 | 12
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypokinesia (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Myoclonic epilepsy (Nervous system disorders) | 1 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0
Petit mal epilepsy (Nervous system disorders) | 1 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0
Somnolence (Nervous system disorders) | 5 | 11 | 7
Tremor (Nervous system disorders) | 0 | 2 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0
Apathy (Psychiatric disorders) | 0 | 1 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Enuresis (Psychiatric disorders) | 0 | 0 | 1
Epileptic psychosis (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 2 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 1
Soliloquy (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Thinking abnormal (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
Lymphocyte morphology abnormal (Investigations) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT01747915/SAP_000.pdf
  • Study Protocol (2012-07-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT01747915/Prot_001.pdf